CLINICAL TRIAL: NCT06742840
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-2129 Following Multiple Doses Administration in Healthy Subjects
Brief Title: A Multiple Ascending Dose Trial of HRS-2129 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2129-102
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-2129 experimental group (Experimental)
  Interventions: Drug: HRS-2129
- HRS-2129 placebo group (Placebo Comparator)
  Interventions: Drug: HRS-2129 placebo

INTERVENTIONS:
Drug: HRS-2129 — HRS-2129.
  Arms: HRS-2129 experimental group
Drug: HRS-2129 placebo — HRS-2129 placebo.
  Arms: HRS-2129 placebo group

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HRS-2129 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 55 years old (inclusive);
2. Body weight: ≥ 50 kg for male and ≥ 45 kg for female, body mass index: 19.0 ~ 28.0 kg/m2 (inclusive);
3. Subject has no plan to give a birth, donate sperm or eggs from signing the informed consent form to 6 months after last dose;
4. Female subjects: non-pregnant or non-lactating;
5. The skin to receive pain stimuli has no wound or derma disease;
6. Subject who is willing to accept pain test;
7. Subject who voluntarily signs the informed consent.

Exclusion Criteria:

1. Subject who suffers from clinical acute and chronic diseases of circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormalities;
2. Subject with a history of torsade de pointes, symptomatic or multigenic or frequent or require medical treatment arrhythmia, or personal or family history of short QT syndrome or long QT syndrome;
3. Subject with a history of allergies to the IMP or its excipients, or subject with allergic constitution;
4. Subject who underwent major surgery within 6 months prior to screening, or received surgery that may significantly affect the pharmacokinetics or safety evaluation of the IMP, or who plans to undergo surgery during the study period;
5. Subject with a medication history that inhibits or induces liver metabolism of drug has been used within 1 month before administration;
6. Subject with vaccinated within 1 month prior to screening or plan to be vaccinated during the study;
7. Subject who used any drugs or health products (including Chinese herbal medicines) within 7 half-lives or 14 days (whichever is longer) before administration, or who plans to receive other drug treatments during the study;
8. Subject who has participated in clinical trials and received experimental drugs within 3 months before screening, or plans to participate in other clinical trials during this study;
9. Donate blood/blood loss ≥ 400 mL within 3 months before screening;
10. Subject who smoked more than 5 cigarettes per day on average within 3 months before screening;
11. Drink more than 14 units of alcohol per week on average;
12. Drink excessive tea, coffee or caffeinated beverages within 3 months before screening;
13. Consume special food (such as grapefruit, grapefruit juice or food/drink containing grapefruit juice, chocolate, tobacco, alcohol, caffeine and other food or drink) within 48 hours before administration;
14. Subject who has special requirements for diet and cannot follow a unified diet;
15. Subject with clinical significant abnormalities in medical examination;
16. Subject with positive tests for hepatitis B surface antigen, hepatitis C virus antibody, syphilis or human immunodeficiency virus antibody;
17. Subject with a history of drug abuse or with a positive result for drug abuse test;
18. Alcohol test result is positive;
19. Subject who has difficulty in swallowing, or venous blood collection, or who cannot tolerate venipuncture, or who has a history of fainting of needle or blood;
20. Subject who is judged to have suicidal ideation or suicidal behavior by mental state assessment;
21. Subject may not be able to complete the study due to other reasons or the investigators considers that he is not suitable for inclusion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AEs) | From ICF signing date to Day 39.
The incidence and severity of adverse events (AEs) | From ICF signing date to Day 41.

SECONDARY OUTCOMES:
Cold Pain detection threshold for the Thermode Cold Test | Day 1 to Day 12.
Cold Pain detection threshold for the Thermode Cold Test | Day 1 to Day 15.
Heat Pain detection threshold for the Thermode Heat Test | Day 1 to Day 12.
Heat Pain detection threshold for the Thermode Heat Test | Day 1 to Day 15.
Pain tolerance time for the Cold Pain Test | Day 1 to Day 12.
Pain tolerance time for the Cold Pain Test | Day 1 to Day 15.
Number of participants with clinically meaningful findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses | From ICF signing date to Day 13.
Number of participants with clinically meaningful findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses | From ICF signing date to Day 15.
Time to reach maximum plasma concentration (Tmax) of HRS-2129 | 0 hour to 216 hours after administration.
Terminal half-life (t1/2) | 0 hour to 216 hours after administration.
Maximum plasma concentration (Cmax) of HRS-2129 | 0 hour to 216 hours after administration.
Apparent clearance (CL/F) of HRS-2129 | 0 hour to 216 hours after administration.
Apparent volume of distribution (Vz/F) of HRS-2129 | 0 hour to 216 hours after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided